CLINICAL TRIAL: NCT07400289
Title: M149 - Development of a FibroScan Liver Examination Using a Single Probe
Brief Title: Development of a FibroScan Liver Examination Using a Single Probe
Acronym: M149
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Collaborators: Novotech CRO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M149
Record Dates: First submitted 2025-12-22; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Liver Diseases
Keywords: FibroScan; Liver stiffness Measurement; Vibration Controlled Transient Elastography
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): Adult patients followed in the Hepatology department for a chronic liver disease, all etiologies combined.
  Interventions: Device: Research FibroScan

INTERVENTIONS:
Device: Research FibroScan — *Patients #1 to #50: Exam 1: Examination with Research FibroScan and single probe #1 (SP1). Exam 2: Examination with Research FibroScan and single probe #2 (SP2). Exam 3: Examination with Research FibroScan and single probe #3 (SP3). Exam 4: Examination with the Reference FibroScan at the same measurement point. The examination must start alternatively with the FS exam using the SP1 probe, the SP2 probe or the SP3 probe to avoid potential bias.
  The standard examination must be always done at the end, after the first 3 exploratory exams.
  *Patients #51 to #309: Exam 1: Examination with the Research FibroScan. Exam 2: Examination with the Reference FibroScan at the same measurement point. The examination must start alternatively with the Research FibroScan and the Reference FibroScan to avoid potential bias.

SUMMARY:
This is an exploratory, international, prospective, interventional, multicenter clinical investigation that will take place in 1 Hong Kong site and 3 French sites and 309 adults patients will be included. The study objective is to assess the LSM reproducibility between the FibroScan examination performed with the Single Probe (SP) and the FibroScan examination performed with the reference probes (M and XL).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years of age).
* Patient followed with a chronic liver disease.
* Adult patient able to give his written consent.
* For European sites: patient affiliated to the healthcare system.

Exclusion Criteria:

* Vulnerable patients.
* Patients with ascites.
* Patients with heart failure.
* Patients with acute hepatitis.
* Patients with biliary obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference between LSM by guided-VCTE performed with the single probe and LSM by guided-VCTE performed with the reference probes (M and XL). | At Day 0
  This outcome assesses the difference between the values of LSM obtained with the single probe and the reference probes (M and XL) when performed in the same patients.

SECONDARY OUTCOMES:
Difference between CAP performed with single probe and CAP performed with the reference probes (M and XL). | At Day 0
  This outcome assesses the difference between the CAP measurements obtained with the single probe and the reference probes (M and XL) when performed in the same patients.
Difference of patient percentage having a successful examination between the FibroScan (guided-VCTE) examination performed with the single probe and the FibroScan (guided-VCTE) examination performed with the reference FibroScan probes (M and XL probes). | At Day 0
  This outcome compare the applicability of FibroScan examinations performed with the single probe compared with the reference probes (M and XL).
Difference between the values reported by the patient on the comfort scale after a FibroScan (guided-VCTE) examination performed with the single probe and after a FibroScan examination (guided-VCTE) performed with the reference probes (M and XL). | At Day 0
  This outcome evaluates the difference in patient-reported comfort following FibroScan examinations performed with the single probe versus the reference probes (M and XL), as reported by patients after undergoing the examinations under similar conditions. A comfort scale from 0 to 10 will be given to the patients, where 10 represents the most confortable and 0 the more incomfortable.

CONTACTS AND LOCATIONS:
Locations (4):
- France (3):
  - CHRU de Besançon, Besançon
  - Hôpital St Eloi- CHU Montpellier, Montpellier
  - Hôpital Paris Saclay, Orsay
- Prince of Wales Hospital the Chinese University of Hong Kong, Hong Kong, Hong Kong